CLINICAL TRIAL: NCT03685656
Title: Randomized, Double-blind, Placebo Controlled Trial of Effect of ANACA3 Slimming Gel on Loss of Abdominal and Thigh Circumferences in Healthy Volunteers
Brief Title: Effect of ANACA3 Slimming Gel on Loss of Abdominal and Thigh Circumferences in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nutravalia (Industry)
Collaborators: Slb Pharma (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: EFFANACA3GEL
Record Dates: First submitted 2018-07-16; First posted 2018-09-26 (Actual); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Overweight and Obesity
Keywords: Overweight; Obesity; Slimming gel; Cosmetic product; Waist circumference; Thigh circumference
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ANACA3 (Experimental): ANACA3 slimming gel
  Interventions: Other: Slimming gel
- Placebo (Placebo Comparator): Slimming gel contening no active ingredient
  Interventions: Other: Slimming gel placebo

INTERVENTIONS:
Other: Slimming gel — On the morning, one application per day on each area under study (thighs and abdomen) during 8 weeks.
  Other Names: ANACA3 Le Gel Minceur
  Arms: ANACA3
Other: Slimming gel placebo — On the morning, one application per day on each area under study (thighs and abdomen) during 8 weeks.
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
Overweight and obesity is defined, according to the World Health Organization (WHO), by abnormal or excessive accumulation of adipose or fatty tissue that may be harmful to health.

Overweight and obesity are therefore important determinants of health, which expose people to many pathologies whose consequences for individuals are not only health, but also social: stigma, prejudice, discrimination.

Indeed, most overweight people have a bad image of themselves. For some people, overweight can trigger stress, malaise and disgust.

To break free from this malaise and satisfy the growing desire of women to take care of their body, many products are present in the slimming beauty market.

EFFANACA3GEL is a prospective, randomized, double-blind, placebo controlled study. 208 healthy volunteers will be followed for 2 months during which they will use ANACA3 slimming gel. The aim of this study is to evaluate the effects of ANACA3 slimming gel on hip and waist circumferences.

ELIGIBILITY:
Inclusion Criteria:

* Healthy woman,
* Age between 18 and 65 years,
* Body mass index (BMI) strictly greater than 23 kg / m² and strictly less than 35 kg / m² with a stable weight (± 2 kg) for at least 3 months,
* Stable physical activity for at least 3 months,
* Lack of firmness in the abdomen and thighs,
* Presenting cellulite visible in the thighs, with a score of 3 to 8 according to the photographic scale used,
* Hormonal treatment not modified for at least 3 months,
* informed and written consent signed.

Exclusion Criteria:

* Pregnant or lactating woman,
* Use of a slimming product and / or anti-cellulite (oral or topical) in the month prior to participating in the study,
* Slimming diet during the last 3 months,
* Special diet: low calorie diet (slimming diet and / or medication taken with or without a significant increase in physical activity over the last 3 months) or special diet (vegetarians, vegans, any intake of nutritional supplements )
* Smoking (more than 3 cigarettes per day) and/ or addiction to alcohol,
* Consuming more than 3 cups of coffee and / or tea per day,
* Active evolutionary pathology or a history of cancer,
* Under corticosteroids or any other medicinal treatment that may have an influence on water retention without therapeutic balance at the time of inclusion,
* Antecedent of surgery for bariatric and / or aesthetic,
* Severe eating disorders (anorexia, bulimia, binge eating, etc.),
* Not affiliated to a Social Security scheme.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 208 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-02-13 (Actual); Study Completion 2019-02-13 (Actual)

PRIMARY OUTCOMES:
Waist circumference | 8 weeks
  Measure of the waist circumference using a measuring tape.

SECONDARY OUTCOMES:
Waist circumference | 2 weeks
  Measure of the waist circumference using a measuring tape.
Abdominal circumference | 2 and 8 weeks
  Measure of the abdominal circumference (at the level of the navel) using a measuring tape.
Hip circumference | 2 and 8 weeks
  Measure of the hip circumference using a measuring tape.
Thigh circumference | 2 and 8 weeks
  Measure of thigh circumference using a measuring tape.
Abdominal skinfold using a Harpenden skinfold caliper | 2 and 8 weeks
  Measure of the abdominal skinfold using a Harpenden skinfold caliper
Cellulite | 2 and 8 weeks
  Scoring of cellulite in the thighs using a photography scale Scale: 8 photographies - Grade 0 to Grade 8; Hiher the grade is, more there is cellulite.
Elasticity and firmness of the abdominal skin | 2 and 8 weeks
  Measure of the elasticity and firmness of the abdominal skin using a cutometer

CONTACTS AND LOCATIONS:
Locations (1):
- GREDECO, Paris, France